CLINICAL TRIAL: NCT00451347
Title: Comparison of The Clinical Effects Between Different Physical Therapy Tools in Patellofemoral Pain Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 200611006R
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2006-11

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

INTERVENTIONS:
Device: Quadriceps strength training
Device: Taping
Device: Home exercise

SUMMARY:
Objectives:The purpose of this study was to investigate the different effects among the quadriceps strength training, taping, and stretching exercise of iliotibial band in patients with patellofemoral pain syndrome by randomized control trial study.

Method:An observer blind, prospective, factorial design randomized controlled trail. 90 young adults with patellofemoral pain syndrome were randomly allocated into one of three treatment groups: (1) Quadriceps strength training, (2) taping, and (3) stretch. Each group received treatment for 8 weeks.

Hypothesis:Patients in quadriceps strength training group may get most outcomes in three groups

DETAILED DESCRIPTION:
Introduction:Patellofemoral pain syndrome ( PFPS ) is a common knee disorder. Factors that cause patellofemoral pain include: over use, soft tissue imbalance, and malalignment of lower extremity. Patients with patellofemoral pain, caused by soft tissue imbalance was thought to be favorite to receive physical therapies. Clinically, physical therapies for patients with PFPS are including: Quadriceps strength training, taping, and stretching exercise. The aforementioned treatment tools showed different effect mechanism. However, there were few clinical studies to compare the clinical effects among the aforementioned three treatment tools. The purpose of this study was to investigate the different effects among the quadriceps strength training, taping, and stretching exercise of iliotibial band in patients with patellofemoral pain syndrome by randomized control trial study.

Methods:An observer blind, prospective, factorial design randomized controlled trail. 90 young adults with patellofemoral pain syndrome were randomly allocated into one of three treatment groups: (1) Quadriceps strength training, (2) taping, and (3) stretch. Each group received treatment for 8 weeks.

Outcome measures were including visual analog scales for worst pain, active-active joint reposition error test, the Chinese version of the Western Ontario and McMaster Universities Osteoarthritis Index, and one repetition maximum recorded at baseline and after the interventions for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Anterior or retropatellar knee pain present during at least two of the following: ascending/descending stairs, hopping, running, squatting, kneeling, and prolong sitting
* Insidious onset of symptom unrelated to a traumatic incident
* Pain on palpation of peripatella
* VAS>3
* Age <50 years old
* Symptoms sustained for more than 1 month

Exclusion Criteria:

* Over activity: athlete, infatry
* Patients with meniscal lesion, ligamentous instability, patellar tendon pathology, radiation pain from spine, referred pain
* Neurological disease involved

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90
Dates: Start 2006-11; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
VAS worst
muscle strength
proprioception
functional performance

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Hwa Jan, Study Director — Kinesiology Lab, School and Graduate Institute of Physical Therapy, National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, National Taiwan University, Taipei, Taiwan